CLINICAL TRIAL: NCT00077545
Title: A Phase II Study Of Triapine In Combination With Cisplatin Esophageal Carcinoma
Brief Title: 3-AP Plus Cisplatin in Treating Patients With Recurrent or Metastatic Adenocarcinoma of the Esophagus or Gastroesophageal Junction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02576; NCI-2012-02576 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000352307; UCCRC-12765A; NCI-6285; 12765A (Other: University of Chicago Comprehensive Cancer Center); 6285 (Other: CTEP); N01CM62201 (NIH)
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Adenocarcinoma of the Esophagus; Recurrent Esophageal Cancer; Stage IV Esophageal Cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms | interventions — 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; Cisplatin

ARMS (1):
- Treatment (triapine and cisplatin) (Experimental): Patients receive 3-AP (Triapine) IV over 2 hours on days 1-4. Patients also receive cisplatin IV over 60 minutes on days 2 and 3 before 3-AP infusion. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: triapine; Drug: cisplatin

INTERVENTIONS:
Drug: triapine — Given IV
Drug: cisplatin — Given IV

SUMMARY:
Drugs used in chemotherapy, such as 3-AP and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. 3-AP may help cisplatin kill more cancer cells by making them more sensitive to the drug. This phase II trial is studying how well giving 3-AP together with cisplatin works in treating patients with recurrent or metastatic adenocarcinoma of the esophagus or gastroesophageal junction.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate in patients with recurrent or metastatic adenocarcinoma of the esophagus or gastroesophageal junction treated with 3-AP (Triapine) and cisplatin.

SECONDARY OBJECTIVES:

I. Determine the toxicity of this regimen in these patients. II. Determine the duration of response and overall survival of patients treated with this regimen.

III. Determine the palliative benefits with regard to dysphagia in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive 3-AP (Triapine) IV over 2 hours on days 1-4. Patients also receive cisplatin IV over 60 minutes on days 2 and 3 before 3-AP infusion. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed for up to 2 years.

PROJECTED ACCRUAL: A total of 19-39 patients will be accrued for this study within 20 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the esophagus or gastroesophageal junction

  * Metastatic or recurrent disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
  * Outside prior irradiation port
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 50-100%
* More than 6 months
* Absolute neutrophil count ≥ 1,500/mm^3
* WBC ≥ 3,000/mm ^3
* Platelet count ≥ 100,000/mm^3
* AST and ALT ≤ 2.5 times upper limit of normal
* Bilirubin normal
* Creatine normal
* Creatinine clearance ≥ 50 mL/min
* No prior myocardial infarction
* No unstable angina
* No cardiac arrhythmia
* No uncontrolled congestive heart failure
* No pulmonary disease requiring supplemental oxygen
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No glucose-6-phosphate dehydrogenase (G6PD) deficiency (for patients of African, Asian, or Mediterranean origin)
* No other concurrent uncontrolled illness
* No active or ongoing infection
* No active second malignancy
* No prior allergic reaction to compounds of similar chemical or biological composition to 3-AP or other study agents
* No psychiatric illness or social situation that would preclude study compliance
* At least 1 year since prior platinum-derivative agents
* No prior chemotherapy for metastatic or recurrent esophageal cancer
* See Disease Characteristics
* At least 2 weeks since prior radiotherapy and recovered
* No other concurrent anticancer therapy
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2004-01; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Complete response rate | Up to 2 years
  Will be calculated together with 95% confidence intervals based on the binomial distribution.
Objective response rate (CR + PR) | Up to 2 years
  Will be calculated together with 95% confidence intervals based on the binomial distribution.

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
  Kaplan-Meier estimates will be determined.
Progression-free survival | From the start of treatment to progression or death, assessed up to 2 years
  Kaplan-Meier estimates will be determined.
Duration of response | From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 2 years
Number of patients with various treatment-related toxicities assessed using NCI CTCAE version 3.0 | Up to 2 years
Number of patients with improvement of dysphagia | Up to 2 years
Duration of improvement of dysphagia | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ann Mauer, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States